CLINICAL TRIAL: NCT01344005
Title: A Pilot Clinical Trial Looking at the Effect on Lung Cancer Diagnosis of Giving a CXR to Smokers Aged Over 60 With Chest Symptoms
Brief Title: Standard Medical Care or Urgent Chest X-ray in Diagnosing Lung Cancer in Smokers With Chest Symptoms Who Are Older Than 60 Years
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wales Cancer Trials Unit (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000699222; WCTU-EL-CID; EU-21112; CRUK-C8350/A12199
Record Dates: First submitted 2011-04-27; First posted 2011-04-28 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2011-04

CONDITIONS: Lung Cancer; Tobacco Use Disorder
Keywords: non-small cell lung cancer; small cell lung cancer; tobacco use disorder
MeSH Terms: conditions — Lung Neoplasms; Tobacco Use Disorder; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — X-Rays

INTERVENTIONS:
Other: caregiver-related intervention or procedure
Other: questionnaire administration
Procedure: quality-of-life assessment
Procedure: radiography

SUMMARY:
RATIONALE: Diagnostic procedures, such as an urgent chest x-ray, may help in planning cancer treatment. It is not yet known whether standard medical care is more effective than an urgent x-ray in diagnosing lung cancer in smokers with chest symptoms who are older than 60 years.

PURPOSE: This randomized clinical trial is studying standard medical care to see how well it works compared with an urgent chest x-ray in diagnosing lung cancer in smokers with chest symptoms who are older than 60 years.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the prevalence of extra-NICE symptoms in patients consulting in UK general practice.
* To determine the proportion of patients who agree to participate in the trial.
* To determine the proportion of patients who are diagnosed with lung cancer and the best sources of routine data for capturing lung cancers.

Secondary

* To determine the best way to train general practitioners to identify and recruit eligible patients into the trial.
* To determine the most effective method of presenting the trial (and randomization) to patients.
* To determine the barriers to recruitment and how to overcome those barriers.
* To determine the best tools to use to measure anxiety/depression that may be caused by unnecessary chest-x-rays or no chest x-rays.
* To determine the best measures of resource use to facilitate health economic analysis of the cost-effectiveness of 'extra-NICE'.
* To determine the stage at diagnosis, performance status, and the proportion of patients receiving radical treatments in those diagnosed with lung cancer.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm A: Patients are managed as per the National Institute for Health and Clinical Excellence (NICE) guidelines.
* Arm B: Patients are referred for an urgent chest x-ray according to extra-NICE guidelines.

General practitioners from South East Wales are surveyed to assess their level of interest in the proposed full trial. For the feasibility study, 20 South East Wales general practices and 6 South Yorkshire general practices are selected. General practitioners are trained to recruit all patients who fulfill the extra-NICE criteria as well as those who do not.

Patients complete questionnaires (HADS, EQ-5D, and ICECAP[O]) at baseline and at 2 months to measure quality of life and health economic analysis of the cost-effectiveness of extra-NICE guidelines.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients over 60 seeing a participating General Practitioner
* Currently smokes 10 or more pack years, meeting at least one of the following criteria:

  * New or altered cough of any duration reported to primary care
  * Increased breathlessness or wheezing (with or without purulent sputum)
* Do not qualify for an urgent referral for a chest x-ray under the National Institute for Health and Clinical Excellence (NICE) guidelines (i.e., hemoptysis or unexplained or persistent [lasting > 3 weeks] signs or symptoms), including having any of the following:

  * Cough
  * Chest/shoulder pain
  * Dyspnea
  * Weight loss
  * Chest signs
  * Hoarseness
  * Finger clubbing
  * Features suggestive of metastasis from a lung cancer (e.g., in the brain, bone, liver, or skin)
  * Cervical/supraclavicular lymphadenopathy

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* No chest x-ray within in past 3 months
* No need for a chest x-ray within the next 3 weeks for reasons other than those listed under Disease Characteristics

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of extra-NICE symptoms in patients consulting in UK general practice
Proportion of patients who agree to participate in the trial
Proportion of patients who are diagnosed with lung cancer and the best sources of routine data for capturing lung cancers

SECONDARY OUTCOMES:
Best way to train general practitioners to identify and recruit eligible patients into the trial
Most effective method of presenting the trial (and randomization) to patients
Barriers to recruitment and how to overcome those barriers
Best tools to use to measure anxiety/depression that may be caused by unnecessary chest-x-rays or no chest x-rays
Best measures of resource use to facilitate health economic analysis of the cost-effectiveness of 'extra-NICE'
Stage at diagnosis, performance status, and the proportion of patients receiving radical treatments in those diagnosed with lung cancer
False-positive and false-negative rates for chest x-rays

CONTACTS AND LOCATIONS:
Overall Officials: Richard Neal, MD, Principal Investigator — North Wales Clinical School

REFERENCES:
- [Derived] Prout H, Tod A, Neal R, Nelson A. Maximising recruitment of research participants into a general practice based randomised controlled trial concerning lung diagnosis-staff insights from an embedded qualitative study. Trials. 2022 Mar 21;23(1):225. doi: 10.1186/s13063-022-06125-y. PMID 35313926
- [Derived] Prout HC, Barham A, Bongard E, Tudor-Edwards R, Griffiths G, Hamilton W, Harrop E, Hood K, Hurt CN, Nelson R, Porter C, Roberts K, Rogers T, Thomas-Jones E, Tod A, Yeo ST, Neal RD, Nelson A. Patient understanding and acceptability of an early lung cancer diagnosis trial: a qualitative study. Trials. 2018 Aug 4;19(1):419. doi: 10.1186/s13063-018-2803-4. PMID 30075741
- [Derived] Neal RD, Barham A, Bongard E, Edwards RT, Fitzgibbon J, Griffiths G, Hamilton W, Hood K, Nelson A, Parker D, Porter C, Prout H, Roberts K, Rogers T, Thomas-Jones E, Tod A, Yeo ST, Hurt CN. Immediate chest X-ray for patients at risk of lung cancer presenting in primary care: randomised controlled feasibility trial. Br J Cancer. 2017 Jan;116(3):293-302. doi: 10.1038/bjc.2016.414. Epub 2017 Jan 10. PMID 28072761
- [Derived] Hurt CN, Roberts K, Rogers TK, Griffiths GO, Hood K, Prout H, Nelson A, Fitzgibbon J, Barham A, Thomas-Jones E, Edwards RT, Yeo ST, Hamilton W, Tod A, Neal RD. A feasibility study examining the effect on lung cancer diagnosis of offering a chest X-ray to higher-risk patients with chest symptoms: protocol for a randomized controlled trial. Trials. 2013 Nov 26;14:405. doi: 10.1186/1745-6215-14-405. PMID 24279296